CLINICAL TRIAL: NCT02713516
Title: Low-Cost, Virtual Reality System to Increase Access to Exposure Therapy for Anxiety and Obsessive Compulsive Disorders
Brief Title: Virtual Reality System to Increase Access to Exposure Therapy for Anxiety and OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen Whiteside, Associate Professor of Psychology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-008235
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Anxiety; Obsessive Compulsive Disorder
Keywords: Anxiety; OCD; Obsessive Compulsive Disorder; Generalized Anxiety; Social Phobia; Separation Anxiety; GAD; Youth; Teen; Therapy
MeSH Terms: conditions — Anxiety Disorders; Obsessive-Compulsive Disorder; Generalized Anxiety Disorder; Phobia, Social; Anxiety, Separation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): The children in this study will have a single visit. During this visit the child and their parent will be introduced to the virtual reality (VR) system. The child will interact with the VR system and after they have finished, they will be asked questions about their experience with the VR system.
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Use of virtual reality to deliver exposure therapy
  Other Names: Google Cardboard

SUMMARY:
Cognitive Behavioral Therapy with fear provoking exposures is the most effective therapy for anxiety disorders. Investigators aim to enhance this therapy with the use of virtual reality exposures and to make therapy more available and accessible for patients with anxiety disorders. The societal benefit of increased access to therapy is that, if successful, it will increase the number of patients who receive appropriate treatment for an anxiety disorder.

DETAILED DESCRIPTION:
Twenty children with CADs or OCD who have received less than 3 treatment sessions and a parent will be recruited to pilot the VR system. Participants will be identified through the Mayo Clinic Pediatric Anxiety Disorders Clinic. Each patient will participate in a single (up to) 2-hour visit. During the first 30 minutes the patient and parent will be introduced to the VR system and the rationale for this feasibility study. Next, a therapist will lead the patient through exposure exercises using the VR system for up to 30 minutes. During the next period, up to 30 minutes, the therapist will go to a different room and the patient, with support from their parent, will complete exposure exercises using the VR system that the therapist directed them to complete. During the exposures the interviewer will observe, code and record the patient's interaction with the VR system. For the remaining time (up to 30 minutes) the interviewer will interview the patient about his or her experience with the VR system and then will ask for observations and opinions from the parent.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7 to 12
2. Primary diagnosis of anxiety, generalized anxiety disorder, social phobia, separation anxiety and/or OCD

Exclusion Criteria:

1. History of and/or current diagnosis of: psychosis, autism, bipolar disorder, mental retardation, oppositional defiant disorder, PTSD, selective mutism or major depressive disorder.
2. Current suicidality or recent suicidal behavior
3. Parent to be involved in study who is unable to adequately participate due to intellectual or psychiatric difficulties
4. Starting or changing the dosage of a psychiatric medication in the last 2 months

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in Subjective Units of Distress Scale (SUDS) at end of session | approximately 2 hours
  The SUDS - 0 to 10 ratings, where 0 indicates that they feel no anxiety at all and 10 indicates that they are experiencing maximum distress

SECONDARY OUTCOMES:
Percent of children to describe the virtual reality system as engaging and easy to use based on qualitative interviews | approximately 2 hours
  The ease of use of the VR system

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Whiteside, PhD., L.P., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
We are collecting user acceptability/feasibility data in a small pilot